CLINICAL TRIAL: NCT02618564
Title: The Use of Sennosides With Pico Salax in Bowel Preparation for Colonoscopy: a Study of Optimal Dose and Timing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DMED#1845-15
Record Dates: First submitted 2015-10-03; First posted 2015-12-01 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Colonoscopy Preparation Outcome
MeSH Terms: interventions — Sennosides

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2 TABS QHS (Active Comparator): Sennosides 2 tabs, taken two nights before the colonoscopy
  Interventions: Drug: Sennosides
- 3 TABS QHS (Active Comparator): Sennosides 3 tabs, taken two nights before the colonoscopy
  Interventions: Drug: Sennosides
- 2 TABS AM (Active Comparator): Sennosides 2 tabs, taken the morning before the colonoscopy
  Interventions: Drug: Sennosides
- 3 TABS AM (Active Comparator): Sennosides 3 tabs, taken the morning before the colonoscopy
  Interventions: Drug: Sennosides
- 2 TABS AM & QHS (Active Comparator): Sennosides 2 tabs taken the morning before and 2 tabs taken the evening before the colonoscopy.
  Interventions: Drug: Sennosides

INTERVENTIONS:
Drug: Sennosides — Each group will be assigned different doses of sennosides and varying times of administration
  Other Names: Senokot

SUMMARY:
The objective of this study is to evaluate sennosides as an adjunct to sodium picosulfate magnesium citrate (Pico Salax) in preparation for colonoscopy. We will compare different doses and administration times. The primary outcome is number of bowel motions produced. Secondary outcomes include the quality of bowel cleansing and patient tolerability.

DETAILED DESCRIPTION:
We will compare different doses and administration times in patients booked for morning colonoscopy. The primary outcome is number of bowel motions produced in total by the sennosides. Secondary outcomes include the quality of bowel cleansing and patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female patients 18 to 75 years of age inclusive
* Patients who require an outpatient colonoscopy with a split dose Pico-Salax prep

Exclusion Criteria:

* Colonoscopy requiring the use of a large volume prep (eg Colyte, PEG)
* Ileus or bowel obstruction
* Previous colorectal surgery
* Ascites
* Recognized renal impairment (defined as GFR less than normal in 3 months prior to enrolment)
* Pregnancy
* Recent (<6 months) myocardial infarction or unstable angina.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Bowel movements, as measured by patient diary | 2 days
  The primary outcome of this pilot study is the number of bowel movements. Patients will record the timing and number of bowel motions produced.

SECONDARY OUTCOMES:
Colon cleansing, as measured by The Ottawa Scale and Aronchick Bowel Cleansing Scale | 2 days
  The secondary outcome is colon cleansing efficacy. The endoscopist will grade the cleansing quality of the colon using two standardized measures - the Ottawa Scale and the 5-point Aronchick Bowel Preparation Scale
Tolerability, as measured by patient questionnaire | 2 days
  The secondary outcome is patient tolerability. Patients will be asked to complete a questionnaire examining symptoms such as nausea, bloating, vomiting, and abdominal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No